CLINICAL TRIAL: NCT05633485
Title: The Effect of Animation-Supported Education Based on the Health Promotion Model for Protection From COVID-19 Disease on Primary School Students
Brief Title: Animation Supported COVID-19 Education
Acronym: COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Siirt University (Other)
Responsible Party: Principal Investigator, Sidar Gül, Principal Investigator, Siirt University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2021-SİÜSBF-032
Record Dates: First submitted 2022-11-29; First posted 2022-12-01 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2022-11

CONDITIONS: COVID-19 Pandemic
Keywords: Animation-Supported Education; COVID-19; School-Age Children; Healthy Life
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): An animation-supported training based on the health promotion model for COVID-19 disease and prevention measures was given to the participants.
  Interventions: Other: Animation-Supported Education
- Control (No Intervention): No intervention was applied to the participants in the control group.

INTERVENTIONS:
Other: Animation-Supported Education — Expert support was received for the design and preparation of animation videos.
  Arms: Experimental

SUMMARY:
Introduction: The COVID-19 epidemic and related mutations, which affect the whole world, continue to increase globally. In particular, this crisis adversely affects school-age children's quality of life.

Method: The study was carried out between February and April 2022 following the experimental research criteria with the pretest-posttest-retest control group. The research population consists of 4th-grade primary school students studying in schools affiliated with the Siirt Directorate of National Education. The sample consists of 148 students studying in the 4th grade at two schools deemed suitable for the conduct of the study. Data were collected using data collection materials, the Descriptive Questionnaire, and the General Child Quality of Life Scale.

Results: The mean age of all students participating in the study was 10.53±2.60, 53% of the students were girls, and 47% were boys. It has been determined that 36.0% of the Students have not received any training on COVID-19 before, 32.4% of them did not take precautions to defend themselves from COVID-19 disease, and it is not possible to protect 48.4% of them from COVID-19 disease even if adequate precautions are taken. It was found that the difference between the pretest, posttest, and retest mean scores of the Students in the experimental group on the quality of life scale was statistically significant (p < 0.05). It was determined that the mean of life quality increased immediately after the training but decreased in the measurements one month later.

Conclusion: Education to be given to school-age children should be developed with animation-supported programs.

DETAILED DESCRIPTION:
The new type of Coronavirus Disease (COVID-19), which emerged in China in December 2019, has spread rapidly worldwide. It was declared a global pandemic by the World Health Organization on March 11, 2020 (WHO, 2020). COVID-19 poses a significant threat to the entire society. For this, educational institutions that seem to be risky among the measures taken worldwide have been closed (1). For this reason, it has been decided to continue all education activities through distance education from November 20, 2020, until January 4, 2021. Afterward, it was decided to conduct face-to-face education and training activities in certain stages (2,3).

The importance of education and information activities to prevent COVID-19 disease and reduce the spread of the disease is indisputable. Due to the initiation of face-to-face education, informing school-age children about prevention from the epidemic plays a crucial role in making the school environment safe (4). One of the methods that can be used to inform school-age children about COVID-19 is animations created within the scope of play therapy because animations provide psychomotor, cognitive, social, and emotional development of children and give them positive behaviors and habits (5-7). Concordantly, nurses who stay in close and long-term communication with children, as are with all segments of society, have tremendous responsibilities. Providing accessible, accurate, and evidence-based health information about the epidemic is among the accountabilities of nurses (8). Benefiting from theories and models that offer a professional approach to nursing has many benefits, such as increasing the quality of education, guiding practice, and increasing the health level of individuals (9). For this purpose, the health promotion model (10), created by Pender is suitable to be used in nursing studies carried out to protect against COVID-19 disease

ELIGIBILITY:
Inclusion Criteria:

* Being at school between the study dates
* Volunteering of the students' and parents' willingness to participate in the research

Exclusion Criteria:

* The presence of a communication problem in the participant

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 148 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Socio-demographic Questionnaire | Baseline
  This form was developed by the researchers in line with the literature and consists of 10 questions. In the form, there are five questions about the students' socio-demographic characteristics and five queries about their knowledge and perceptions of the COVID-19 disease.
Generic Quality of Life Instrument for Children (Kid-KINDL) | Baseline
  The questionnaire consists of 6 subscales; Physical state, psychological well-being, self-worth, family, friend, and school subscales. The scale consists of 30 items in a 5-point Likert type. High scores indicate a healthy quality of life.
Generic Quality of Life Instrument for Children (Kid-KINDL) | At the end of the 1st week
  The questionnaire consists of 6 subscales; Physical state, psychological well-being, self-worth, family, friend, and school subscales. The scale consists of 30 items in a 5-point Likert type. High scores indicate a healthy quality of life.
Generic Quality of Life Instrument for Children (Kid-KINDL) | At the end of the 4th week
  The questionnaire consists of 6 subscales; Physical state, psychological well-being, self-worth, family, friend, and school subscales. The scale consists of 30 items in a 5-point Likert type. High scores indicate a healthy quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Siirt University, Siirt, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No